CLINICAL TRIAL: NCT02659553
Title: Impact of Graft Steatosis on Post-operative Complications After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Collaborators: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Emad Ali Ahmed Ali, Principal Investigator, Sohag University
Other Study IDs: 28/9/2014
Record Dates: First submitted 2016-01-11; First posted 2016-01-20 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Post-operative Complications
Keywords: Liver Transplantation - Steatosis - Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- mild steatosis: 5% - 30% of hepatocytes have fatty infiltration
  Interventions: Procedure: steatosis
- moderate steatosis: 30% - 60% of hepatocytes have fatty infiltration
  Interventions: Procedure: steatosis
- No steatosis: No or less than 5% of hepatocytes have fatty infiltration
  Interventions: Procedure: steatosis

INTERVENTIONS:
Procedure: steatosis — Liver Transplantation with graft steatosis

SUMMARY:
1. Clinical impact of graft steatosis on postoperative complications after OLT.
2. Recommendations to improve outcomes after transplantation of steatotic livers and increase donor pool.

DETAILED DESCRIPTION:
Introduction Solid organ transplantation has become the standard of care for selected patients with end-stage organ dysfunction. With improved surgical techniques, more effective immunosuppressive therapies, and better anti-infective medications, outcomes after solid organ transplantation have improved over the last several years.

The excellent survival rates reported after orthotopic liver transplantation (OLT) have increased the demand for liver transplants and have enhanced the disparity between the number of available donor organs and the need for such organs.

The lack of available organs for liver transplantation (LT) associated with the increased death rates among patients on most waiting lists for LT has triggered the use of so-called extended criteria donor (ECD) grafts, previously called ''suboptimal grafts''. Among the wide range of these ECD livers, hepatic steatosis is one of the most frequent disorders, which is mostly related to an increasing prevalence of non-alcoholic fatty liver disease (NAFLD).

Non-alcoholic fatty liver disease (NAFLD) is increasingly significant in healthy individuals for its high worldwide prevalence, an association with the metabolic syndrome such as insulin resistance, diabetes, dyslipidemia and obesity, and an association with liver-related morbidity and mortality.

Clinical evaluation and current imaging modalities, and serological and laboratory tests can be strongly suggestive of the presence of hepatic steatosis, but none of these is capable of distinguishing steatohepatitis (SH) from uncomplicated steatosis; likewise, these evaluations can generally detect advanced liver disease (e.g. portal hypertension), but none can truly assess the degree of liver necroinflammatory injury, lesser stages of fibrosis and architectural remodeling. Liver biopsy evaluation, therefore, remains the 'gold standard' to unequivocally diagnose SH and to document the severity of hepatic injury and fibrosis.

Steatosis is assessed according to the pattern and the amount of fatty infiltration in hepatic tissue sections. Traditionally, fatty accumulation has been classified morphologically as macrovesicular or microvesicular. Macrovesicular steatosis is characterized by a single, bulky fat vacuole in the hepatocyte that displaces the nucleus to the edge of the cell. The less conspicuous microvesicular steatosis, usually related to toxins or metabolic disorders, is characterized by accumulation of tiny lipid vesicles in the cytoplasm of hepatocytes without nuclear dislocation. Current quantification and grading of liver steatosis originates from studies performed in the early 1990s, when steatosis was classified as mild, moderate, or severe if, less than 30%, 30-60%, or more than 60% of hepatocytes, respectively, display fatty infiltrations.

Although usually benign, fatty liver may associate with serious injury, with inflammation and hepatocyte necro-apoptosis, non-alcoholic steatohepatitis (NASH), in 20-30% of subjects. Those patients are at risk of developing fibrosis, one fifth progressing to liver cirrhosis. It is apparently more slowly progressive than other chronic liver diseases, such as alcohol or viral-induced disease. Moreover, the problem of hepatocytes being fatty, overcomes the liver itself, as it increases the risk for cardiovascular disease and death and duplicates the risk for type 2 diabetes mellitus (T2DM), independently of the severity of liver injury.

Severe fatty livers are more susceptible to warm and cold ischemia reperfusion injury than normal ones. The type of damage is not through the pathway of cellular apoptosis, but necrosis.

The use of steatotic grafts for orthotopic liver transplantation (OLT) is associated with a high rate of primary graft dysfunction and decreased graft and patient survival particularly with macro-steatosis.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients candidates for liver transplantation are included in this study

Exclusion Criteria:

* Pediatric patients are excluded.
* Re- transplanted patients.
* cases with no histopathological examination records

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients candidate for liver transplantation are included in this study
Sampling Method: Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Post-operative complications rate | through study completion, an average of 1 year
  according to the Clavien- Dindo classification system

SECONDARY OUTCOMES:
Biliary complications: stricture or leakage | through study completion, an average of 1 year
  the outcome will be measured retrospectively from the hospital records and prospectively in the recent cases of transplantation
early graft dysfunction (EGD), which is defined as impaired initial allograft function with high peak serum transaminase and persistent high bilirubin levels. | through study completion, an average of 1 year
  the outcome will be measured retrospectively from the hospital records and prospectively in the recent cases of transplantation
Primary graft non-function (PNF), which is defined as primary failure of the graft followed by death or re-transplantation within the first post transplantation week. | through study completion, an average of 1 year
  the outcome will be measured retrospectively from the hospital records and prospectively in the recent cases of transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Alaa A. Redwan, Professor, Study Director — Sohag University; Marco Vivarelli, Professor, Study Director — Università Politecnica delle Marche
Locations (1):
- Polytechnic university of Marche, Ancona, AN, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nocito A, El-Badry AM, Clavien PA. When is steatosis too much for transplantation? J Hepatol. 2006 Oct;45(4):494-9. doi: 10.1016/j.jhep.2006.07.017. Epub 2006 Jul 31. No abstract available. PMID 16919359
- [Result] El-Badry AM, Jang JH, Elsherbiny A, Contaldo C, Tian Y, Raptis DA, Laczko E, Moritz W, Graf R, Clavien PA. Chemical composition of hepatic lipids mediates reperfusion injury of the macrosteatotic mouse liver through thromboxane A(2). J Hepatol. 2011 Dec;55(6):1291-9. doi: 10.1016/j.jhep.2011.04.019. Epub 2011 May 19. PMID 21703192
- [Result] Trevisani F, Colantoni A, Caraceni P, Van Thiel DH. The use of donor fatty liver for liver transplantation: a challenge or a quagmire? J Hepatol. 1996 Jan;24(1):114-21. doi: 10.1016/s0168-8278(96)80195-4. No abstract available. PMID 8834034
- [Result] Lee JY, Kim KM, Lee SG, Yu E, Lim YS, Lee HC, Chung YH, Lee YS, Suh DJ. Prevalence and risk factors of non-alcoholic fatty liver disease in potential living liver donors in Korea: a review of 589 consecutive liver biopsies in a single center. J Hepatol. 2007 Aug;47(2):239-44. doi: 10.1016/j.jhep.2007.02.007. Epub 2007 Mar 6. PMID 17400323
- [Result] McCormack L, Dutkowski P, El-Badry AM, Clavien PA. Liver transplantation using fatty livers: always feasible? J Hepatol. 2011 May;54(5):1055-62. doi: 10.1016/j.jhep.2010.11.004. Epub 2010 Nov 13. PMID 21145846
- [Result] Machado MV, Cortez-Pinto H. Non-invasive diagnosis of non-alcoholic fatty liver disease. A critical appraisal. J Hepatol. 2013 May;58(5):1007-19. doi: 10.1016/j.jhep.2012.11.021. Epub 2012 Nov 23. PMID 23183525